CLINICAL TRIAL: NCT04366986
Title: International Registry of Coronavirus Exposure in Pregnancy (IRCEP)
Brief Title: International Registry of Coronavirus (COVID-19) Exposure in Pregnancy
Acronym: IRCEP
Status: Completed | Type: Observational
Sponsor: Pregistry (Industry)
Collaborators: Harvard School of Public Health (HSPH) (Other)
Responsible Party: Sponsor
Other Study IDs: 0001
Record Dates: First submitted 2020-04-23; First posted 2020-04-29 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Covid-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pregnant Women: Women who are currently pregnant
  Interventions: Other: Tested for SARS-CoV-2 (regardless of the result); Other: Clinical diagnosis of COVID-19 by a health care professional
- Post-partum women: Women who have been pregnant in the past 6 months
  Interventions: Other: Tested for SARS-CoV-2 (regardless of the result); Other: Clinical diagnosis of COVID-19 by a health care professional

INTERVENTIONS:
Other: Tested for SARS-CoV-2 (regardless of the result) — This is an observational study with no intervention
Other: Clinical diagnosis of COVID-19 by a health care professional — This is an observational study with no intervention

SUMMARY:
The International Registry of Coronavirus Exposure in Pregnancy (IRCEP) is a prospective cohort study of pregnant and recently pregnant women who have been tested for SARS-CoV-2 (regardless of the result) or have been clinically diagnosed with COVID-19 by a health care professional. Data from the IRCEP will be used to evaluate the impact of COVID-19 on pregnancy and birth outcomes.

DETAILED DESCRIPTION:
The International Registry of Coronavirus Exposure in Pregnancy (IRCEP) will enroll women 18 years of age and older who are currently pregnant or have been pregnant women within the last 6 months, and who have been tested for SARS-CoV-2 (regardless of the result) or have been clinically diagnosed with COVID-19 by a health care professional. As this is an international registry, women from all countries are welcome to participate.

Women will enroll and provide information to the IRCEP via website and mobile app. After signing the electronic informed consent document, registrants will answer questions on the following modules: Demographics, Reproductive History, Height and Weight, Habits, Health Conditions, Medications, Current Pregnancy, COVID-19 Infection Test, and COVID-19 Infection Symptoms. Monthly follow-up modules will continue until the pregnancy outcome. In case of a live birth, the Registry participant will continue with the Post-Partum Outcomes module until the newborn is 90 days of age. Medical records from the mother and neonate will also be requested.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women or women who have been pregnant within the last 6 months
* Able to give electronic informed consent
* Tested for SARS-CoV-2 (regardless of the result) or clinically diagnosed with COVID-19 by a health care professional

Exclusion Criteria:

* <18 years of age

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Persons assigned gender female at birth.
Study Population: Pregnant women, or women who have been pregnant in the last 6 months, who were tested for SARS-CoV-2 (regardless of the result) or were clinically diagnosed with COVID-19 by a health care professional.
Sampling Method: Non-Probability Sample
Enrollment: 17318 (Actual)
Dates: Start 2020-06-23 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Pregnancy outcomes | 1 year
  Miscarriage (or spontaneous abortion), Elective termination, Stillbirth, Preterm delivery
Birth outcomes | Birth to 90 days post-partum
  Major structural defects, neonatal death, Admission into the Neonatal Intensive Care Unit, Maternal obstetric complications, Post-partum health
Birth outcomes | Birth to 90 days post-partum
  Head circumference at birth in centimeters
Birth outcomes | Birth to 90 days post-partum
  Length at birth in centimeters

CONTACTS AND LOCATIONS:
Overall Officials: Diego Wyszynski, MD, MHS, PhD, Principal Investigator — CEO Pregistry
Locations (1):
- Pregistry, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: International Registry of Coronavirus (COVID-19) Exposure in Pregnancy — https://ircep.pregistry.com